CLINICAL TRIAL: NCT04609670
Title: A Phase 1, Open-Label Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of a Single Oral Dose of [14C]-ALXN2050 in Healthy Adult Male Subjects
Brief Title: Study of Radiolabeled ALXN2050 in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN2050-HV-106
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: Mass Balance; ALXN2050; Factor D Inhibitor; Total Radioactivity; Absorption; Metabolism; Excretion
MeSH Terms: interventions — rhoA GTP-Binding Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-ALXN2050 (Experimental): Participants will receive [14C]-ALXN2050.
  Interventions: Drug: [14C]-ALXN2050

INTERVENTIONS:
Drug: [14C]-ALXN2050 — A single dose of 200 milligrams (~85 microcuries) [14C]-ALXN2050 will be administered orally.
  Other Names: ALXN2050; ACH-0145228 (formerly)

SUMMARY:
This is an open-label study to assess the absorption, metabolism, excretion, and mass balance of a single oral dose of carbon-14 ([14C])-ALXN2050 in healthy adult males.

ELIGIBILITY:
Inclusion Criteria:

1. No clinically significant medical history, physical or neurological examination findings, screening clinical laboratory profiles, or electrocardiogram findings.
2. Body mass index in the range of 18.0 to 32.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50.0 kg at screening.
3. Non-sterile participants must agree to abstinence or use a highly effective method of contraception.

Exclusion Criteria:

1. History of any medical or psychiatric condition or disease that might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
2. History or presence of drug or alcohol abuse within previous 2 years, current user of tobacco/any nicotine-containing product, or positive drugs-of-abuse screen or alcohol screen at screening or Day -1 of Period 1.
3. History or presence of seizures, head injury, or head trauma.
4. History of procedures that could alter absorption or excretion of orally administered drugs.
5. History of meningococcal infection, or has a first-degree relative with a history of meningococcal infection.
6. Body temperature ≥ 38.0°Celcius at screening or check-in.
7. Donation of whole blood from 3 months prior to first dosing or of plasma from 30 days before first dosing, or receipt of blood products within 6 months prior to first dosing.
8. Has less than 1 bowel movement every 2 days or has a recent history of abnormal bowel movements, such as diarrhea, loose stools, or constipation, within 2 weeks prior to dosing.
9. Has received radiolabeled substances or has been exposed to radiation sources within 12 months of dosing or is likely to receive radiation exposure or radioisotopes within 12 months of dosing such that participation in this study would increase their total exposure beyond the recommended levels considered safe.
10. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days prior to dosing, whichever is longer.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Mass Balance Recovery In Urine And Feces After a Single Oral Dose Of [14C]-ALXN2050 | Up to 168 hours postdose or maximum of 504 hours for extended collection period postdose
  Mass balance will be assessed by evaluating total radioactivity recovery and the percent of the radioactive dose excreted in the urine and feces. Mass balance will be calculated as a sum of the percent of the total radioactivity recovered in urine and feces plus any radioactivity dose lost due to emesis (if any occurred) relative to the administered radioactivity dose.
Plasma Pharmacokinetics (PK) Of Total Radioactivity After A Single Oral Dose Of [14C]-ALXN2050: Area Under The Concentration-time Curve From Time 0 Extrapolated To Infinity (AUC0-inf) | Up to 168 hours postdose or maximum of 504 hours for extended collection period postdose
Plasma PK Of Total Radioactivity After A Single Oral Dose Of [14C]-ALXN2050: Area Under The Concentration Versus Time Curve, From Time 0 To The Time Of The Last Measurable Concentration (AUC0-last) | Up to 168 hours postdose or maximum of 504 hours for extended collection period postdose
Plasma PK Of Total Radioactivity After A Single Oral Dose Of [14C]-ALXN2050: Maximum Observed Plasma Concentration (Cmax) | Up to 168 hours postdose or maximum of 504 hours for extended collection period postdose
Plasma PK Of Total Radioactivity After A Single Oral Dose Of [14C]-ALXN2050: Time To Maximum Observed Plasma Concentration (Tmax) | Up to 168 hours postdose or maximum of 504 hours for extended collection period postdose
Plasma PK Of ALXN2050 After A Single Oral Dose Of [14C]-ALXN2050: AUC0-inf | Up to 168 hours postdose
Plasma PK Of ALXN2050 After A Single Oral Dose Of [14C]-ALXN2050: AUC0-last | Up to 168 hours postdose
Plasma PK Of ALXN2050 After A Single Oral Dose Of [14C]-ALXN2050: Cmax | Up to 168 hours postdose
Plasma PK Of ALXN2050 After A Single Oral Dose Of [14C]-ALXN2050: Tmax | Up to 168 hours postdose
Percentage Of Total Radioactivity Detected For Each ALXN2050 Metabolite in Plasma, Urine, And Feces | Up to 168 hours postdose or maximum of 504 hours for extended collection period postdose
  ALXN2050 metabolic profiling in plasma, urine, and feces will be performed in samples containing sufficient amounts of radioactivity. The percent of dose represented by each of the metabolites will be calculated using the radioactivity concentration equivalent data combined with the metabolic profiling data. The percentage of each identified metabolite to total radioactivity in plasma will be estimated based on plasma metabolic profiling data.

SECONDARY OUTCOMES:
Number Of Participants Receiving A Single Oral Administration Of [14C]-ALXN2050 With Treatment-emergent Adverse Events | Day 1 (after dosing) through follow-up (30 [+/- 2] days after dosing on Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No